CLINICAL TRIAL: NCT04749758
Title: Assessment of the Functional, Clinical and Radiological Efficacy of Stromal Vascular Fraction Treatment for Knee Osteoarthritis
Brief Title: Assessment of the Efficacy of Stromal Vascular Fraction Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Andorra (Other)
Responsible Party: Principal Investigator, Anna BOADA-PLADELLORENS, Principal Investigator, University of Andorra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UA003GRCSSS
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; regenerative medicine; mesenchymal stem cells; stromal vascular fraction
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: One-year prospective observational study of patients treated with stromal vascular fraction treatment for knee osteoarthritis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF treatment (Experimental): SVF treatment is developed by Cellab Laboratory (Celstem®). It is approved by Andorra's Government authorities.
  Interventions: Biological: SVF treatment

INTERVENTIONS:
Biological: SVF treatment — SVF treatment is developed by Cellab Laboratory (Celstem®). It is made following strict manufacturing guidelines and approved by Andorra's Government authorities. An abdominal fat liposuction is required to obtained Celstem®. The preparation of the product is carried out exclusively in a clean laboratory room under the conditions described by the AABB (American Association of Blood Banks) standards. The treatments application is carried out on the same day of the extraction, at some point between the next 6 hours from the end of the extraction. Firstly, ultrasound joint evaluation is performed. Under sterility measures, intraarticular infiltration of SVF treatment is performed at affected knee or knees. Previous synovial fluid aspiration is performed, if required. Once the procedure is completed, rehabilitation recommendations and clinical follow-up information is provided.

SUMMARY:
One-year follow-up prospective observational study involving male and female patients (over 18-years-old) with unilateral or bilateral knee osteoarthritis treated with intraarticular injection of stromal vascular fraction (SVF) treatment. Clinical, biological and radiological data before the treatment and 1-month, 6-month and a year after are collected.

The research hypothesis supports that SVF treatment enhance functionality and quality of live, relieves pain and improves magnetic resonance images of joint cartilage in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The research consists on one-year follow-up prospective observational study. It involves male and female patients (over 18-years-old) with unilateral or bilateral knee osteoarthritis treated with intraarticular injection of stromal vascular fraction (SVF) treatment developed by Cellab Laboratory (Celstem®).

The aim of the study is to assess pain efficacy with SVF treatment for knee osteoarthritis patients. To assess pain, Visual Analogue Scale (VAS) is used.

Secondarily, the study aims to determine the differences pre-post treatment with SVF of the secondary outcomes measures: functionality, quality of life and disability. Is is used KOOS scale, Short Form-36 questionnaire (SF-36) and World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) to assess such measures, respectively. It also aims to describe and evaluate the regeneration of joint cartilage of each individual by systematic comparison of magnetic resonance imaging (MRI) before and one year after SVF treatment, measured by Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scale. Moreover, specific sociodemographic and clinical factors that can predict or influence the therapeutic effects and its correlation to biological data (cellularity, immunophenotype, colony formation potency and sterility) will be identified. Adverse events or side effects related to the treatment will be reported.

Both primary and secondary outcome measures are evaluated prior to treatment, at 1-month, 6-months and one year after treatment except for the assessment of disability and the radiological features of the articular cartilage, which are performed only before and one year after. The radiological assessment according to MOCART classification is performed by a radiologist. This specialised physician is not aware of patients evolution in order to obtain minimize subjective bias. In addition, SVF product biological data, such as the amount of sample of extracted adipose tissue, effective dose, cellularity, immunophenotype, potency sample colonies and sterility, are collected to better describe the product and to be able to correlate the clinical effect with biological features.

The study was approved by the Clinical Research Ethics Committee of Nostra Senyora de Meritxell Hospital on September 20th, 2018. It is expected to last 4 years, from 2018 to 2022.

The sample size is determined using the Sample Size Calculator GRANMO (Version 7.12. April 2012). A random sample of 77 individuals affected of knee osteoarthritis is expected to be sufficient to estimate, with 95% confidence and accuracy of +/- 5 percentage units, a population percentage that is expected to be around 5% in the study population (population of the regions of Andorra and Catalonia). A required replacement rate of 5% is expected.

Once treatment indication is been performed and accepted by the patient, patients who meet the inclusion criteria (see Eligible Criteria) sign the informed consent. Personal data transfer consent to medical team is also signed.

Patients can be withdrawn if they do not complete the questionnaires in pre-established time and form or if its tracking is lost. Withdrawal of the patient does not represent any prejudice to the patient in the control of his disease or in its treat by the medical team or the Laboratory.

For clinical data collection, patient's medical history and physical examination, are collected by the principal investigator (PI) or collaborators in every follow-up medical visits. For a better patient compliance with the study protocol, a web platform has been developed (https://www.cellab.com/escalas-de-dolor). It has been designed by PI aided by an external computer team. It allows the virtual patient performance of functional scales all along the study protocol. This tool dumps all data entered by patients into an Excel database, which can be exported for statistical analysis by PI. In addition, the platform warns every time a patient is supposed to fill the questionnaires or even when they do not comply in time and / or form established.

Despite being an observational study, the object under study is a specific treatment of regenerative medicine: SVF treatment developed by Cellab Laboratory (Celstem®). The main feature of this treatment is that it raises the importance of this study is that the product used is made following strict guidelines manufacturing that ensure its reproducibility, quality and safety. It is approved by the Andorra Government authorities for its application.

It should be noted that the procedure for obtaining, preparing and applying Celstem® it is always performed by the same professionals: a plastic surgeon, biotechnologist and a physical medicine and rehabilitation physician (who appears to be the PI), respectively, in order to avoid interpersonal biases in the process.

Obtaining Celstem® requires abdominal fat liposuction. It is performed by a plastic surgeon underneath sedation and local anesthesia in an operating room, under the supervision of a anesthetist. The amount adipose tissue extracted varies according to availability in each patient, with a minimum extraction of 200ml. The extracted tissue is immediately transported (within 1 hour) to Cellab Laboratory in standardized refrigeration conditions. A traceability certificate is filled to ensure its conservation.

The product's preparation is carried out exclusively in a laboratory cleanroom, following American Association of Blood Banks (AABB) standards conditions of hygiene and biological safety. It requires an exhaustive washing of the fat extracted with saline solution in order to remove both residues of blood or lidocaine and adrenaline used in the extraction process. Then the fat is concentrated and mixed with the enzymatic digestion solution (consisting of collagenase at 0.75 mg / mL). It is all incubated at 37 °C and stirred for 30-40 minutes. When this process is finished, collagenase is inactivated through human albumin and then again thoroughly washed with saline solution to remove the remnants of undigested fat and collagenase. A concentrated cell suspension in a reduced volume is obtained.

Once ready, the product returns at the clinic, again under proper refrigeration conditions and with the certificate of traceability correctly complimented to ensure its proper conservation. The application of the treatment is carried out on the same day of the extraction, in some point within 6 hours after the extraction. Under sterility measures, intraarticular infiltration of SVF treatment (Celstem®) is performed at affected knee or knees. Previous synovial fluid aspiration is performed, if required. Once the procedure is completed, rehabilitation recommendations and clinical follow-up information is provided.

ELIGIBILITY:
Inclusion Criteria:

Male and female over 18 years of age patients affected from unilateral or bilateral symptomatic knee osteoarthritis (KOA), determined by the diagnostic criteria of the American College of Rheumatology. Any degree of the Kellgren and Lawrence classification for KOA is included. Patients included must have KOA symptoms more than 6 months. Symptomatology must remain despite having done conventional treatment for KOA.

Exclusion Criteria:

* Suspicion, diagnosis or history of active or recent joint infection (less than 6 months)
* Neurological deficit in the affected limb
* Pregnant or breastfeeding women
* Positive serology for hepatitis B, hepatitis C and / or HIV
* Magnetic resonance imaging without pathological alterations
* Knee infiltration with glucocorticoids, hyaluronic acid, platelet - rich plasma and / or other regenerative medicine therapies in the last 3 months.
* Medical conditions, including the diagnosis of oncological pathology or infectious and severe heart, kidney or liver disease, which contraindicate sedation or liposuction procedure.
* History or diagnosis of dementia or higher functions unpreserved, which interfere communication.
* Not having the necessary skills and / or electronic devices necessary (even their relatives or acquaintances, or they can not help them) to complete the online questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline knee pain measured with a Visual Analogue Scale (VAS) at 1 year | Pain is assessed pre-intervention and at one year of follow-up.
  Joint pain measured using the Visual Analogue Scale (VAS), which allows the patient to score from 0 to 10, 0 being that there is no pain, and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Change from baseline functionality measured with Knee Injury and Osteoarthritis Outcome Score (KOOS) at 1 year | Functionality is assessed pre-intervention and at one year of follow-up.
  Measured by Knee Injury and Osteoarthritis Outcome Score (KOOS). This patient-administered questionnaire consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A total score has not been validated and is not recommended.
Change from baseline quality of life measured with SF-36 questionnaire at 1 year. | Quality of life is assessed pre-intervention and at one year of follow-up.
  Measured using the SF-36 questionnaire. This questionnaire consists of a battery of questions answered in about 10 minutes in order to quantify the general health status of patients. It uses 8 scales to measure three aspects: functional state, well-being and overall subjective assessment of one's own health. 8 numbers are obtained from 0 to 100, taking into account that higher scores mean better health.
Change from baseline disability measured with WHODAS 2.0 questionnaire at 1 year. | Disability is assessed pre-intervention and at one year of follow-up.
  Measured using the 12-item WHODAS 2.0 questionnaire (http://www.who.int/classifications/icf/whodasii/en/). This questionnaire includes 12 items out of 6 disability domains contemplating 2 components (activities, which includes cognition, mobility, and self-care; and participation, which includes relationship with third parties, activities of daily living and social participation) during the 30s previous days. Each of the 12 items is scored from 0 to 4, where 0 is assumed no, 1 mild, 2 moderate, 3 severe and 4 extreme or complete difficulty in the specific activity. The total score of the questionnaire ranges from 0 to 48, where the lower, the better the functionality, with 1-4 being a disability mild; 5-9 moderate disability and 10-48 severe disability.
Change from baseline joint cartilage characteristics measured with Magnetic Resonance Imaging at 1 year. | Joint cartilage characteristics are assessed pre-intervention and at one year of follow-up.
  Measured by magnetic resonance imaging (MRI) following the bases of the MOCART classification (Magnetic Resonance Observation of Cartilage Repair Tissue). This classification scores the thickness, the joint surface, resonance signal and subchondral bone status in each of the three knee joints and the presence or absence of joint spill. It scores 20 points for the normal thickness, 15 if there is hypertrophy, 10 if cartilage is decreased more than 50%, 10 if cartilage is decreased less than 50%.10 points are obtained for the regularity of the surface, 5 if the irregularity exceeds 50% and 0 if it is less than 50%. The score total is between 0 and 55, where higher score means greater alteration of cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Boada-Pladellorens, MD, Principal Investigator — Hospital Nostra Senyora de Meritxell; Mercè Avellanet, PhD, Study Chair — Hospital Nostra Senyora de Meritxell; Esther Pages, PhD, Study Chair — Hospital Nostra Senyora de Meritxell; Josep A Farras Roca, MD, Study Chair — Cente mèdic d'especialitats Dr. Farras
Locations (1):
- CelularClinic, Les Escaldes, Andorra

IPD SHARING:
Plan to Share IPD: No
Study data will not be used by any other researcher.